CLINICAL TRIAL: NCT06629649
Title: Implementing AI-based Glaucoma Screening Within Federally Qualified Health Centers
Acronym: AI-RONA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); University of California, San Diego (Other)
Responsible Party: Principal Investigator, Cynthia Owsley, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Screening
Other Study IDs: IRB-300013425; 1U01DP006827-01 (NIH)
Record Dates: First submitted 2024-09-30; First posted 2024-10-08 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Glaucoma; Ocular Hypertension
Keywords: visual acuity impairment; glaucoma; ocular hypertension; glaucoma suspect; diabetic retinopathy; cataract
MeSH Terms: conditions — Glaucoma; Ocular Hypertension; Diabetic Retinopathy; Cataract | interventions — Mass Screening

STUDY DESIGN:
Intervention Model Description: The initial design implements the eye screening intervention in 4 FHQC clinics operated by Southeast Alabama Rural Health Associates (SARHA) for a duration of 18 months. Four other FQHC clinics operated by SARHA are the control, or non-interventional clinics, which are followed during the same time period. After 18 months the control clinics become the interventional clinics and the previous intervention clinics become the control clinics.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The Federally Qualified Health Centers (FQHCs) (Experimental): Eight FQHCs will participate in this project. Four FQHCs will implement a glaucoma screening protocol and a protocol for detecting diabetic retinopathy, cataract, and visual acuity impairment, while the other four will be standard of care without the above screening protocol.
  Interventions: Other: Glaucoma screening using an AI-algorithm and screening for diabetic retinopathy, cataract, and visual acuity impairment.
- Primary Standard of Care (No Intervention): Primary care provider asks participants if they are having symptoms or problems with their eyes or vision.

INTERVENTIONS:
Other: Glaucoma screening using an AI-algorithm and screening for diabetic retinopathy, cataract, and visual acuity impairment. — Participants who have the glaucoma screening will undergo an Artificial Intelligence Remote Optic Nerve Assessment (AI-RONA). The AI information may or may not be used by the FQHC provider to refer their patient for follow-up eye exam. It is information that the provider may find useful in making a referral.
  Arms: The Federally Qualified Health Centers (FQHCs)

SUMMARY:
The goal of this clinical trial is to learn if implementation of an eye screening program at Federally Qualified Health Center (FQHC) clinics provides results that participants may have glaucoma, and/or other eye conditions (diabetic retinopathy, cataract, visual acuity impairment). The glaucoma screening will incorporate use of an artificial intelligence (AI)-assisted screening tool. This project is called AI-RONA. The main questions it aims to answer are:

* How does this eye screening program compare to the rate of glaucoma and other eye conditions detected at other FQHC clinics where the screening program has not been implemented?
* Do particpants who screen positive for these conditions adhere to the physician's recommendation for a follow-up examination by an optometrist or ophthalmologist?
* Are referral rates for a follow-up comprehensive eye exam by an optometrist or ophthalmologist similar to those implemented by an ophthalmologist using telemedicine (that is, using the results of the screening to make a diagnosis remotely)?
* What is the cost-effectiveness of the AI-assisted screening program in diagnosing glaucoma as compared to a physician-guided program?
* Are participants completing the screening satisfied with it?
* Are physicians at the FQHC clinics administering the screening satisfied with it?

Participants will:

* Undergo an ocular screening whose goal is to detect glaucoma, diabetic retinopathy, cataract, and/or impairment in visual acuity. If the screening indicates that participants may have these conditions, participants will be referred for a comprehensive eye examination by an optometrist or ophthalmologist.
* Following the screening, participants and physicians will complete a survey on their satisfaction with the program.

DETAILED DESCRIPTION:
Federally Qualified Health Center (FQHC) clinics are excellent candidate clinics for eye disease screening programs for adults, including glaucoma and also other glaucoma associated diseases (GAD), diabetic retinopathy, cataract and refractive error. These clinics are safety-net primary health care clinics in the United States designed to serve medically underserved areas and populations. The physician will provide services regardless of the patient's ability to pay, using a sliding-scale fee based on the ability to pay. Over half the patient population at FQHCs nationally is Black or Hispanic, with 82% of patients uninsured or federally insured. While FQHCs provide primary medical care in many health domains, one domain that is not adequately addressed by FQHC clinics is eye care. A recent report by the National Academies of Science, Engineering and Medicine indicated that primary eye care services (through optometrists or ophthalmologists) are rarely available at FQHC clinics; the report provided an estimate that less than 3% of FQHC patients actually receive vision care services at these clinics, representing 0.89% of FQHC clinic visits.

The screening methods used in this protocol are a modified version of our prior imaging-based ophthalmologist guided telemedicine screening protocol utilized in the previous CDC- funded Alabama Screening and Intervention for Glaucoma and eye Health through Telemedicine (AL-SIGHT) study. In AL-SIGHT we used a telemedicine program to screen for glaucoma in 3 FQHCs located in a low-income, under-resourced region of the state with a high proportion of Black residents. Just as we did in AL-SIGHT, investigators in the current protocol will target screening only for those FQHC patients at-risk for glaucoma. The eligibility definition for screening in the current project is listed under Eligibility.

After screening, patients with a screening diagnosis of GAD, diabetic retinopathy, cataract, or visual acuity impairment will be referred for an in-person follow-up exam by an ophthalmologist or optometrist located in the FQHC clinic's region. In the investigators' previous project, participants had excellent adherence to the follow-up appointment with the optometrist or ophthalmology at a rate of 76.7% of patients attending follow-up. Thus, Investigators are hopeful that in the current project they will also have this high level of adherence.

There are two major differences between our previous project (AL-SIGHT) and the current project AI-RONA. In AL-SIGHT, we used research staff members to do the screening at the FQHCs. In AI-RONA investigators will now use implementation science to do the screening. This means that investigators will train the FQHC clinic staff to do the screening after a detailed training and certification program. A second way AI-RONA differs from AL-SIGHT is that investigators will use an AI-assisted, remote screening algorithm to generate the screening results for glaucoma. Investigators will also focus on both the effectiveness of the program (disease detection, rate of referrals) and primary care providers (PCPs) and patients' attitudes about AI-RONA. The latter will be achieved by administering a questionnaire to PCPs and to participants about their satisfaction with the screening program.

The AI approaches to be deployed for AI-RONA have been previously developed and extensively tested by the AI-researchers at the University of California, San Diego, who are also investigators in AI-RONA. It was found that glaucoma testing using AI based on retinal images taken of patients' eyes lead to clinician-level accuracy. These AI methodologies have been tested on diverse populations and publicly available datasets to facilitate their accuracy.

The eye screen protocol that investigators are using includes the following. All assessments are performed on each eye separately: (1) retinal imaging including fundus photography and optical coherence tomography (OCT), (2) visual acuity measurement, (3) refractive error measurement.

ELIGIBILITY:
Inclusion Criteria:

* African American or Hispanic persons ≥ 40 years old
* Non-Hispanic white persons ≥ 50 years old
* Anyone ≥ 18 years old with diabetes type 1 or type 2
* Anyone ≥ 18 years old who already has a glaucoma associated disease
* Anyone ≥ 18 years old with a family history of glaucoma

Exclusion Criteria:

* Declines to sign written informed consent
* Cannot communicate in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1800 (Estimated)
Dates: Start 2025-10-22 (Actual); Primary Completion 2029-09-29 (Estimated); Study Completion 2029-09-29 (Estimated)

PRIMARY OUTCOMES:
Rate of participants where the glaucoma screening protocol leads to a screening diagnosis of glaucoma | up to 2-3 days
  Primary care provider will make a screening diagnosis of glaucoma associated disease based on the results of the screening
Rate of participants who decide to attend the follow up exam by optometrist or ophthalmologist | up to 4 months
  If diagnosed with any of the above conditions, and primary car provider recommends follow-up care with an optometrist or ophthalmologist, whether participant actually attends the exam
Rate of participants where the screening protocol leads to a screening diagnosis of cataract, diabetic retinopathy, or visual acuity impairment | up to 2-3 days
  Based on results of screening, the primary care provider will be able to make a screening diagnosis of cataract, diabetic retinopathy or visual acuity impairment
Compare cost of screening program in FQHC to the cost of an ophthalmologist or optometrist guided assessment | up to 4 years
  Compare the cost of AI based interventions relying on optic disc photos alone, OCT alone, both imaging modalities, and imaging with standard vision tests performed by an ophthalmologist or optometrist guided program

SECONDARY OUTCOMES:
Rate of primary care provider who state they agree with intervention acceptability, appropriateness, and feasibility | up to 6 months
  Whether the primary care provider agrees with the eye screening program per the Acceptability of Intervention Measure, Intervention Appropriateness Measure, and Feasibility of Intervention Measure; scores range from 16 to 80 with higher scores meaning more agreement
Rate of participants who state they agree with the acceptability of the screening intervention | up to 1 day
  Whether the participant agrees with the acceptability of eye screening per Post AI-RONA Screening questionnaire; scores range from 9 to 45 with higher scores meaning more agreement

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Owsley, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- Department of Ophthalmology and Visual Sciences, University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Yes
de-identified data will be shared.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: September 29, 2029
Access Criteria: Scientists who work in the field of glaucoma screening and other types of eye screening will be able to access the supporting information described above. They can access this information by contacting the principal investigator.
URL: https://www.uab.edu/medicine/ophthalmology/faculty/owsley